CLINICAL TRIAL: NCT04902976
Title: Evaluation of Viral Load of SARS-COV-2 Virus in the Oral Cavity After Rinsing With Oral Antimicrobial Mouthwashes in Patients Covid-19.
Brief Title: Evaluation of SARS-COV-2 Viral Load of Covid-19 Patients After Rinsing With Oral Antimicrobial Mouthwashes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 4560-21
Record Dates: First submitted 2021-05-24; First posted 2021-05-26 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2021-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — cytidylyl-(3'-5')-cytidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CPC+Zn (Active Comparator): patients submitted to mouth rinse with 0.075% Cetylpyridinium Chloride associated with 0.28% zinc lactate solution.
  Interventions: Other: CPC+ZN
- CPC (Active Comparator): patients submitted to mouth rinse with 0.075% Cetylpyridinium Chloride solution.
  Interventions: Other: CPC
- Negative Control (Placebo Comparator): patients submitted to mouth rinse with distilled water.
  Interventions: Other: Negative Control

INTERVENTIONS:
Other: CPC+ZN — In patients hospitalized in common beds, and without mechanical ventilation, the it will be asked to perform the following procedures: mouth rinse with 20 mL of the solution for 30 s
  Arms: CPC+Zn
Other: CPC — In patients hospitalized in common beds, and without mechanical ventilation, the it will be asked to perform the following procedures: mouth rinse with 20 mL of the proposed solution for 30 s;
  Arms: CPC
Other: Negative Control — In patients hospitalized in common beds, and without mechanical ventilation, the it will be asked to perform the following procedures: mouth rinse with 20 mL of distilled water for 30 s.
  Arms: Negative Control

SUMMARY:
The aim of this study is to analyze the efficacy of oral disinfection with 0.075% Cetylpyridinium Chloride alone and 0.075% Cetylpyridinium Chloride associated with 0.28% zinc lactate in reduction of the viral load of SARS-CoV-2 in the oral cavity. Patients of both sexes, in the age-range between 18 and 90 years, diagnosed positive for SARS-CoV-2 by the RT-PCR method, and who demand oral hygiene care and other preventive and therapeutic dental procedures, will be included in this randomized clinical study.The study will comprise patients hospitalized in common beds, without mechanical ventilation - who will be divided into three groups. Some of these protocols with the use of antimicrobial solutions are hoped to be efficient in reducing the viral load in the oral cavity. This is a factor that could contribute to reducing contamination of the environment caused by aerosols resulting from dental procedures, in addition to helping with the improvement in biosafety protocols against SARS-CoV-2.

DETAILED DESCRIPTION:
Each group of patients will receive specific interventions, as follows: 0.075% Cetylpyridinium Chloride mouthwash (Group 1); 0.075% Cetylpyridinium Chloride associated with 0.28% zinc lactate mouthwash (Group 2), negative control, distilled water (Group 3). To monitor the viral load, the following procedures will be performed: saliva collection, in time intervals before mouth rinsing with the solutions at baseline (T0), immediately after (T1), 30 min (T2), and 1 hour after mouth rinses (T3). SARS-CoV-2 will be quantified by Real Time quantitative reverse transcription polymerase chain reaction (RT-qPCR) assays.

ELIGIBILITY:
Inclusion Criteria:

* positive for SARS-CoV-2 by the RT-PCR method,
* in common bed for minimum of 1 day and maximum of 5 days,
* ensuring that patients are no more than 10 days since showing the first symptoms,
* who are positive for SARS-CoV-2 in the first collection of oral fluid and saliva, and
* who demands oral hygiene care and other preventive and therapeutic dental procedures.

Exclusion Criteria:

* pediatric patients, t
* hose who tested negative for SARS-CoV-2 by the RT-PCR method at the time of recruitment or at the time of first oral fluid and saliva collection;
* those who exhibit oral ulcerations and other erosive lesions in the oral mucosa, which contraindicate the use of cetylpyridinium;
* patients who have bleeding in the oral cavity which prevents sample collections; patients who report history of allergy, irritations or other side effects derived from the use of these substances;
* patients who do not adhere to oral care protocols or those in whom it was not possible to perform these procedures.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-04-04 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Change of SARS-COV-2 load in the oral cavity and saliva | 1 hour
  Change of SARS-COV-2 load in the oral cavity and saliva mensuared by virus fold reduction and viral quantitation

CONTACTS AND LOCATIONS:
Overall Officials: luciana Correa, PhD, Study Director — University of Sao Paulo; Debora H Douek, PhD, Study Chair — Hospital Israelita Albert Einstein
Locations (1):
- Hospital israelita Albert Einstein, São Paulo, Brazil